CLINICAL TRIAL: NCT00268047
Title: Retrospective Assessment of Pulmonary Vascular Resistance in Fontan Patients Who Have Undergone Orthotopic Heart Transplantation
Brief Title: Pulmonary Resistance in Fontan Who Have Undergone Heart Transplantation
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Kirk R Kanter, MD, Children's Healthcare of Atlanta
Other Study IDs: 03-068
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; surgery; transplantation; pulmonary vascular resistance in Fontan patients
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Clinical evidence reveals that some patients who undergo cardiac transplantation exhibit problems with pulmonary vascular resistance as well. In some studies, an increase in pulmonary vascular resistance has been used as an indicator for increased 3-day and 3-month mortality after heart transplantation2. In this study, the investigators would like to look at pulmonary vascular resistance in patients with a surgical history of the Fontan procedure followed by heart transplantation.

DETAILED DESCRIPTION:
Children born with certain congenital heart diseases such as tricuspid atresia or single ventricle physiology normally undergo the Fontan procedure during their course of treatment. The Fontan procedure however is palliative and some of these children will eventually require heart transplantation. It has been shown in pre-clinical animal models that pulmonary vascular resistance actually increases after having the Fontan procedure however this has not been quantitated in the human population.1

This is a retrospective chart review with the primary objective of examining Fontan patients with pulmonary vascular resistance and who have undergone heart transplantation. We will review 50 charts at Children's Healthcare of Atlanta, Egleston Hospital. Three other United States' sites are participating. All de-identified data will be forwarded to the Great Ormond Street Hospital in London, England for study analysis. In order to ascertain this objective, the following data will be collected.

1. Diagnosis
2. Surgical History
3. Information from Pre-transplant evaluation
4. Post-transplant hemodynamics
5. Post-transplant catheterization results

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone the Fontan procedure
* patients cared for at Children's Healthcare of Atlanta
* Patients who have undergone a heart transplantation at Children's Healthcare of Atlanta

Exclusion Criteria:

* Those patients who do meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: retro chart review
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R. Kanter, MD, Principal Investigator — Emory Univ. SOM Cardiothoracic Surgery at Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States